CLINICAL TRIAL: NCT04558060
Title: Randomized, Controlled Evaluation of a Virtual Human Patient for Provider Training in Motivational Interviewing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Greg Reger, Deputy Associate Chief of Staff, VA Puget Sound Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: DM150015
Record Dates: First submitted 2020-09-08; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Motivational Interviewing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Motivational interviewing skill is coded by assessors blind to training condition and assessment time point.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Standardized Patient (Experimental): Training for 45 minutes at each training time point with a computer program that presented a virtual human patient and two simulated patient encounters. The virtual standardized patient involves a branching story line. Participants select 1 of 3 computer-generated response options at each conversational pause: 1) a response that is consistent with the principles and skills of MI, 2) an MI inconsistent response, or 3) a response that is mixed - partly consistent and partly inconsistent with MI.
  Interventions: Other: Virtual Standardized Patient
- Academic Study (Active Comparator): Study of a summary handout of motivational interviewing concepts and techniques for 45-minutes.
  Interventions: Other: Academic Study

INTERVENTIONS:
Other: Virtual Standardized Patient — Computer program that presented a virtual human patient
  Arms: Virtual Standardized Patient
Other: Academic Study — Study of a summary of motivational interviewing concepts and techniques.
  Arms: Academic Study

SUMMARY:
The purpose of this study is to evaluate the efficacy of training with a virtual standardized patient on the acquisition and maintenance of motivational interviewing skills compared with traditional academic study.

DETAILED DESCRIPTION:
Motivational interviewing is an evidence-based counseling approach that aims to increase a patient's motivation to make positive health changes in their lives. A common training method for medical professionals is the use of human standardized patients, who are actors who pretend to be patients for educational interviews. Standardized patients are expensive and it is challenging to maintain an adequate pool of patient actors. Accordingly, after licensure or medical boards, health professionals typically adopt new evidence-based practices, like motivational interviewing, without human standardized patient training experiences. Given the established importance of post-training coaching and feedback to the acquisition of motivational interviewing, innovative training methods are needed. Computer virtual patients may provide a cost-effective alternative that is scalable and supports dissemination of evidence-based practices. This study will evaluate the efficacy of a virtual standardized patient, relative to academic study, for training motivational interviewing among health care professionals from the Department of Veterans Affairs and Department of Defense.

ELIGIBILITY:
Inclusion Criteria:

* All health care staff (e.g., physicians, nurses, social workers, psychologists) from supporting service lines are eligible to participate in the study.

Exclusion Criteria:

* 8 hours or more of formal training in MI in the year prior to baseline assessment.
* Successfully completed participation in the VA Evidence Based Practice roll-out of MI.
* Served as MI trainers or have conducted research on MI at any time
* Do not anticipate being available for the full duration of the training study (according to their verbal self-report)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2016-10-17 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Difference in Motivational Interviewing Treatment Integrity 4.2.1 between the conditions | Change in Motivational Interviewing Treatment Integrity 4.2.1 from Baseline to post-training [approximately 2-weeks after baseline]
  The Motivational Interviewing Treatment Integrity 4.2.1 is a behavioral coding system for motivational interviewing (MI) skill that involves observer ratings of 4 items on a 5-point Likert-type scale and behavior counts. The 5-point scores for Cultivating Change Talk and Softening Sustain Talk are averaged for a Technical Global summary score, and 5-point scores for Partnership and Empathy are averaged for a Relational Global summary score. Behavior counts include simple reflections, complex reflections and questions posed to patients. These behavior counts generate 2 summary scores; the percentage of reflections that are complex reflections and the ratio of reflections to questions. Participants are also categorized as meeting 'fair' and 'good' MI skill proficiency cut points for each of the 4 summary scores.
Difference in Motivational Interviewing Treatment Integrity 4.2.1 between the conditions | Change in Motivational Interviewing Treatment Integrity 4.2.1 from Baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  The Motivational Interviewing Treatment Integrity 4.2.1 is a behavioral coding system for motivational interviewing (MI) skill that involves observer ratings of 4 items on a 5-point Likert-type scale and behavior counts. The 5-point scores for Cultivating Change Talk and Softening Sustain Talk are averaged for a Technical Global summary score, and 5-point scores for Partnership and Empathy are averaged for a Relational Global summary score. Behavior counts include simple reflections, complex reflections and questions posed to patients. These behavior counts generate 2 summary scores; the percentage of reflections that are complex reflections and the ratio of reflections to questions. Participants are also categorized as meeting 'fair' and 'good' MI skill proficiency cut points for each of the 4 summary scores.
Difference in Motivational Interviewing Treatment Integrity 4.2.1 between the conditions | Change in Motivational Interviewing Treatment Integrity 4.2.1 from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  The Motivational Interviewing Treatment Integrity 4.2.1 is a behavioral coding system for motivational interviewing (MI) skill that involves observer ratings of 4 items on a 5-point Likert-type scale and behavior counts. The 5-point scores for Cultivating Change Talk and Softening Sustain Talk are averaged for a Technical Global summary score, and 5-point scores for Partnership and Empathy are averaged for a Relational Global summary score. Behavior counts include simple reflections, complex reflections and questions posed to patients. These behavior counts generate 2 summary scores; the percentage of reflections that are complex reflections and the ratio of reflections to questions. Participants are also categorized as meeting 'fair' and 'good' MI skill proficiency cut points for each of the 4 summary scores.

SECONDARY OUTCOMES:
Difference in Helpful Responses Questionnaire between the conditions | Change in Helpful Responses Questionnaire from Baseline to post-training [approximately 2-weeks after baseline]
  Open-response questionnaire measuring reflective listening skills. Six paragraphs representing discrete things people with a problem might say are presented and participants are asked to write the next thing they would say if they wanted to be helpful. Written responses are coded for the complexity of reflective listening.
Difference in Helpful Responses Questionnaire between the conditions | Change in Helpful Responses Questionnaire from Baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  Open-response questionnaire measuring reflective listening skills. Six paragraphs representing discrete things people with a problem might say are presented and participants are asked to write the next thing they would say if they wanted to be helpful. Written responses are coded for the complexity of reflective listening.
Difference in Helpful Responses Questionnaire between the conditions | Change in Helpful Responses Questionnaire from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  Open-response questionnaire measuring reflective listening skills. Six paragraphs representing discrete things people with a problem might say are presented and participants are asked to write the next thing they would say if they wanted to be helpful. Written responses are coded for the complexity of reflective listening.
Difference in Motivational Interviewing Self-efficacy Scale between the conditions | Change in Motivational Interviewing Self-efficacy Scale from Baseline to post-training [approximately 2-weeks after baseline]
  14-item self-report measure of motivational interviewing self-efficacy
Difference in Motivational Interviewing Self-efficacy Scale between the conditions | Change in Motivational Interviewing Self-efficacy Scale from Baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  14-item self-report measure of motivational interviewing self-efficacy
Difference in Motivational Interviewing Self-efficacy Scale between the conditions | Change in Motivational Interviewing Self-efficacy Scale from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  14-item self-report measure of motivational interviewing self-efficacy
Difference in Provider Knowledge, Skills, and Confidence Survey between the conditions | Change in Provider Knowledge, Skills, and Confidence Survey from baseline to post-training [approximately 2-weeks after baseline]
  Self-reported 3-item measure of MI working knowledge, skills and confidence
Difference in Provider Knowledge, Skills, and Confidence Survey between the conditions | Change in Provider Knowledge, Skills, and Confidence Survey from baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  Self-reported 3-item measure of MI working knowledge, skills and confidence
Difference in Provider Knowledge, Skills, and Confidence Survey between the conditions | Change in Provider Knowledge, Skills, and Confidence Survey from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  Self-reported 3-item measure of MI working knowledge, skills and confidence
Difference in Motivational Interviewing Knowledge and Attitudes Test between the conditions | Change in Motivational Interviewing Knowledge and Attitudes Test from baseline to post-training [approximately 2-weeks after baseline]
  Objective, 14-item test of motivational interviewing knowledge. The measure concludes with a list of MI consistent, inconsistent, or neutral statements and the participant is asked to identify the correct MI principles.
Difference in Motivational Interviewing Knowledge and Attitudes Test between the conditions | Change in Motivational Interviewing Knowledge and Attitudes Test from baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  Objective, 14-item test of motivational interviewing knowledge. The measure concludes with a list of MI consistent, inconsistent, or neutral statements and the participant is asked to identify the correct MI principles.
Difference in Motivational Interviewing Knowledge and Attitudes Test between the conditions | Change in Motivational Interviewing Knowledge and Attitudes Test from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  Objective, 14-item test of motivational interviewing knowledge. The measure concludes with a list of MI consistent, inconsistent, or neutral statements and the participant is asked to identify the correct MI principles.
Difference in Motivational Knowledge Test-Revised between the conditions | Change in Motivational Knowledge Test-Revised from baseline to post-training [approximately 2-weeks after baseline]
  Objective, 18-item multiple choice test of motivational interviewing knowledge
Difference in Motivational Knowledge Test-Revised between the conditions | Change in Motivational Knowledge Test-Revised from baseline to 3-month follow-up training [approximately 3.5-months after baseline]
  Objective, 18-item multiple choice test of motivational interviewing knowledge
Difference in Motivational Knowledge Test-Revised between the conditions | Change in Motivational Knowledge Test-Revised from post-training [approximately 2-weeks after baseline] to 3-month follow-up training [approximately 3.5-months after baseline]
  Objective, 18-item multiple choice test of motivational interviewing knowledge
Difference in Provider Training Satisfaction Survey between the conditions | Post-training [approximately 2-weeks after baseline]
  An 11-item satisfaction survey that assesses participants' satisfaction with the training provided and the degree to which the training enhanced their abilities and preparedness to use MI.

CONTACTS AND LOCATIONS:
Overall Officials: Greg Reger, PhD, Principal Investigator — VA Puget Sound Health Care System

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reger GM, Norr AM, Rizzo AS, Sylvers P, Peltan J, Fischer D, Trimmer M, Porter S, Gant P, Baer JS. Virtual Standardized Patients vs Academic Training for Learning Motivational Interviewing Skills in the US Department of Veterans Affairs and the US Military: A Randomized Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2017348. doi: 10.1001/jamanetworkopen.2020.17348. PMID 33057643